CLINICAL TRIAL: NCT06690710
Title: First-in-human Study to Assess the Safety and Feasibility of Intra-articular Administration of Allogeneic Engineered Gingival Fibroblasts (aeGF) in Patients With Knee Osteoarthritis
Brief Title: FiH Safety and Feasibility Study Assessing Intra-articular Administration of aeGF in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Scarcell Therapeutics S.A.S. (Industry)
Collaborators: TFS Trial Form Support (Industry); Boston Imaging Core Lab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GF-OA-001
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: phase 1; osteoarthritis; knee; cell therapy; ATMP; Advanced Therapy Medicinal Product; Gingival Fibroblasts
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: First in Human, single (expected therapeutic) dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogeneic engineered Gingival Fibroblasts (aeGF), 50 million cells (Experimental): A single intra-articular (IA) injection of 50 million aeGF into one osteoarthritic knee
  Interventions: Biological: allogeneic engineered Gingival Fibroblasts (aeGF)

INTERVENTIONS:
Biological: allogeneic engineered Gingival Fibroblasts (aeGF) — single intra-articular injection of the study drug (aeGF) in the knee joint

SUMMARY:
The company funding this study has developed an advanced therapy medicinal product (a cell therapy) from human donor cells which it wants to assess as a possible treatment for knee osteoarthritis (OA). Tissue from the gums of a human donor is used to make the study drug called allogeneic engineered Gingival Fibroblasts (aeGF). The purpose of this study is to evaluate the safety of a single injection of aeGF in the knee joint of participants with OA. aeGF have shown anti-inflammatory effects, pain relief and cartilage regeneration in animals and so are now being investigated as a treatment for OA in humans.

DETAILED DESCRIPTION:
Scarcell Therapeutics SAS, has developed an advanced therapy medicinal product (a cell therapy) from human donor cells which will be assessed as a possible treatment for knee Osteoarthritis.

Tissue from the gums of a human donor is used to make the study drug called allogeneic engineered Gingival Fibroblasts (from now on aeGF). aeGF are defined as a Tissue Engineered Product (TEPs). TEPs contain cells or tissues that have been modified so that they can repair, regenerate or replace human tissue.

Preclinical studies have been completed which have shown promise in treating osteoarthritis in experimental animal models and domestic animals presenting with osteoarthritis. This study is intended to assess the safety of aeGF in humans for the first time.

In total 15 patients will be dosed with one intra-articular injection of aeGF into the knee, under ultrasound guidance .

The study duration is one year after the injection. A screening visit will take place prior to injection. Eligible participants will return for treatment with the study drug. Followed by a phone call post injection, up to a week later, to assess safety and any side effects of the injection. Hospital follow up visits will occur at 1, 3, 6, 12 and 24 months post injection.

ELIGIBILITY:
Inclusion criteria:

1. Willing and able to provide informed consent;
2. Male or female participants aged ≥40 years;
3. Evidence of OA in the medial tibiofemoral joint (MTJ) as follows:

   * Clinical - knee pain;
   * Radiological - Kellgren-Lawrence:

     1. Grade 2 - definite osteophytes, possible joint space narrowing (JSN), or;
     2. Grade 3 - moderate osteophytes, definite JSN, some sclerosis, possible bone-end deformity (Altman et al., 1986; Kellgren et al., 1957; Kohn et al., 2016).
     3. Minimal joint space width (JSW) of 2.5 mm on knee X-ray (OARSI 1 or 2);
4. Score ≥3 on visual analogue scale (VAS) (0-10 range) for pain at Screening.

Exclusion Criteria:

1. Grade 0, 1 or 4 on the Kellgren-Lawrence grading scale for the target knee:

   * Grade 0: No osteophyte or JSN;
   * Grade 1: Doubtful JSN and possible osteophytic lipping;
   * Grade 4: Large osteophytes, 'bone-on-bone' JSN, severe sclerosis, and definite deformity of bone ends;
2. Severe malalignment of >10° varus or valgus.
3. OA secondary to joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, joint infection, haemophilia, haemochromatosis, calcium pyrophosphate deposition disease, neuropathic arthropathy, trauma, rheumatoid arthritis, gout, psoriatic arthritis, autoimmune arthritis or spondylitis;
4. Receipt of any investigational medicinal product (IMP) or any experimental therapeutic procedure in the 3 months or 5 half-lives before Screening, whichever is longer;
5. Taking corticosteroids or any immunosuppressants, e.g., cyclosporine, prior to Screening;
6. IA treatment with steroids or hyaluronic acid derivatives in the 3 months before Day 1;
7. Planned major surgery, e.g., joint replacement, within 2 months after IA injection;
8. Previous surgery on the target knee including diagnostic arthroscopy;
9. Lesions at the planned injection site that would present a contraindication to local injection of the study drug, e.g., open wounds, psoriatic lesions or infections of the skin;
10. Any known active infection;
11. Clinically significant abnormal haematology or biochemistry values (platelets, haemoglobin, white blood cells, alkaline phosphatase, AST, ALT, blood creatinine, bilirubin) or coagulation (PT, PTT) at Screening;
12. Positive result for HTLV, HIV, Hepatitis B or C;
13. Hypersensitivity to any of the IMP components or excipients;
14. History of sarcoma;
15. History of cancer within five years, except treated basal cell and squamous cell carcinoma of the skin;
16. Women of child-bearing potential, i.e., not post-menopausal (see Section 8.4.5)
17. Women who are pregnant or breastfeeding;
18. Current drug or alcohol abuse;
19. Contraindication to receiving a gadolinium contrast-enhanced magnetic resonance imaging (MRI) of the target knee (metallic implants, claustrophobia, previous anaphylactic reaction to gadolinium, eGFR1 <30 mL/min/1.73 m2, acutely deteriorating renal function) or is unwilling to have MRI performed;
20. Participants with subchondral insufficiency fracture, osteonecrosis, acute or subacute fracture, acute bone contusion, pathologic fracture, stress fracture, fragmentation of articular bone, bone or soft tissue tumour, bone marrow infiltration, posterior meniscal root tear, rheumatoid arthritis, gout based on X-ray or MRI reading;
21. Participants who, in the Investigator's opinion, are unsuitable or unlikely to comply with the study procedures.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
The safety of a single IA injection of aeGF assessed by treatment-emergent adverse events (TEAEs) at 3 months | At 3 months
  A TEAE is defined as an AE observed after starting administration of IMP. The incidence (number and percentage) of participants reporting TEAEs within 3 months after study drug administration will be tabulated. Summaries will be presented by System Organ Class (SOC) and Preferred Term (PT), and further by severity and relationship to IMP.

SECONDARY OUTCOMES:
Change in knee pain and function as assessed by KOOS questionnaire | 1, 3, 6, 12 and 24 months assessments will be compared with baseline
  KOOS is a self-reported patient outcome measure used to assess pain, function, quality of life, and ADL. 42 items are grouped into 5 subscales, i.e.: pain; other symptoms; function in daily living (ADL); Function in Sport and Recreation (Sport/Rec); and, knee-related quality of life. The subscales are scored separately; each yields a score between 0 and 100, with 0 representing extreme knee problems and 100 representing absence of problems. Total KOOS score is the average of all 5 subscale scores; ranging from 0 to 100; where 0 represents extreme knee problems and 100 represents absence of knee problems.
Change in cartilage thickness as assessed by quantitative MRI | Assessed at 12 months and compared with baseline
  Cartilage change will be assessed using the semi-quantitative MRI Osteoarthritis Knee Score (MOAKS) system which is a two-digit score of area size and percentage of subregion affected by full thickness cartilage loss. MOAKS scores articular cartilage in 14 subregions across the knee in 2 dimensions: area of loss as % of subregion surface (AREA); and % of subregion that has full-thickness loss (FTL). AREA and FTL are scored as 0: None; 1: < 10%; 2: 10-75%; 3: >75%.
Change from baseline in biomarker CRP levels | Results at 1, 3 and 12 months will be compared with baseline
  Blood samples will be collected for biomarker, i.e. CRP analysis. CRP will be measured using a standard assay per local laboratory practice.
Use of rescue analgesic medication | Rescue analgesic use at Day 2 and Months 1, 3, 6, 12 and 24 compared with baseline.
  Recording of rescue medication
Change in inflammation as assessed by Contrast-Enhanced Magnetic Resonance Imaging (CE-MRI) | At 6 months and compared with baseline
  Change will be assessed through a contrast enhanced MRI evaluation measuring the level of synovitis in the knee-joint. Inflammation will be measured on an 11-point synovitis score; a reduction by 2 points indicates an improvement.
Incidence, relatedness, severity and duration of TEAEs at 24 months | At 24 months
  The safety of aeGF will be defined by incidence, relatedness, severity and duration of TEAEs at 24 months. The incidence (number and percentage) of participants reporting TEAEs within 24 months after study drug administration will be tabulated. Summaries will be presented by System Organ Class (SOC) and Preferred Term (PT), and further by severity and relationship to IMP.

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust (Nuffield Orthopaedic Centre, Oxford), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No